CLINICAL TRIAL: NCT02339194
Title: Application of a Simplified Method of Complete Denture Fabrication for Severely Resorbed Mandibular Ridges
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal do Ceara (Other)
Collaborators: Fundação Cearense de Apoio ao Desenvolvimento Científico e Tecnológico (Unknown)
Responsible Party: Principal Investigator, Romulo Rocha Regis, Prof. Dr. Rômulo Rocha Regis, Universidade Federal do Ceara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 136958818
Record Dates: First submitted 2015-01-12; First posted 2015-01-15 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Edentulous Mouth; Edentulous Jaw
Keywords: complete denture; quality of life; patient satisfaction
MeSH Terms: conditions — Mouth, Edentulous; Jaw, Edentulous; Patient Satisfaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simplified protocol (Experimental): The application of a simplified denture fabrication technique will be tested for patients presenting severely resorbed mandibular alveolar bones according to the following steps:
  1. Obtainment of maxillary and mandibular casts by using irreversible hydrocolloid in stainless steel stock trays for record bases fabrication.
  2. Adjustment of record bases according to vertical dimension and centric relation measurements, with no use of facebow transfer. Casts will be mounted in semi-adjustable articulator using standardized measures and artificial teeth will be selected.
  3. Trial dentures will be evaluated for esthetics and maxillomandibular relationship.
  4. Insertion of finished dentures.
  Interventions: Procedure: Denture fabrication technique
- Traditional protocol (No Intervention): The importance of a second impression for denture fabrication technique will be tested for patients presenting severely resorbed mandibular alveolar bones according to the following steps:
  1. Maxillary and mandibular casts obtained by using irreversible hydrocolloid in stainless steel stock trays for maxillary record base and mandibular custom tray fabrication.
  2. Mandibular second impression with border molding using compound and impression rubber in custom tray.
  3. Record bases adjustments without facebow transfer. Casts will be mounted in semi-adjustable articulator using standardized measures and artificial teeth will be selected.
  4. Trial dentures will be evaluated for esthetics and maxillomandibular relationship.
  5. Finished dentures insertion.

INTERVENTIONS:
Procedure: Denture fabrication technique — Both arm groups are composed by patients present severely resorbed mandibular alveolar bones who will receive complete dentures fabricated by means of a simpler techinique previously proved to be effective. Although for the "traditional protocol" group a second more complex impression step will be performed in order to evaluate if the simpler approach for this anatomical condition could be safely applied.
  Other Names: Fabrication of complete dentures; Complete denture fabrication technique
  Arms: Simplified protocol

SUMMARY:
BACKGROUND: The literature has shown that simplified methods for complete denture fabrication can be as effective as the traditional techniques, but with less expenditure of time and resources, without prejudice to the patients. However, the effectiveness of these simplified methods for patients with more complex medical conditions haven't been deeply explored.

OBJECTIVES: To evaluate the effectiveness of a proposed simplified method for complete dentures fabrication for patients with severely resorbed mandibular alveolar bones.

METHOD: edentulous patients requesting treatment with bimaxillary complete dentures in a university clinic will be rehabilitated following a simplified technical proposal, being divided randomly into two groups according to the mandibular arch molding technique. In group A, a single impression with alginate through pre-fabricated trays will be performed, while patients allocated in group B will receive a second molding with a more complex technique. After 3 and 6 months, besides important clinical parameters, it will be investigated aspects related to patient's perceptions about the success of treatment. The study will be conducted with a minimum of 30 participants per group, and comparisons between the two groups will be made by means of tests suitable for distribution of data.

ELIGIBILITY:
Inclusion Criteria:

* complete edentulism for at least one year;
* desire to receive a pair of new conventional complete dentures
* mental receptiveness;
* good understanding of spoken Portuguese

Exclusion Criteria:

* disorders of the masticatory system;
* pathological changes of residual ridges;
* debilitating systemic diseases.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Oral health related quality of life | 6 months
  This outcome will be assessed by means of the brazilian version of Oral Health Impact Profile for Edentulous Patients inventory

SECONDARY OUTCOMES:
Satisfaction with dentures (assessed by means of two specific questionaries) | 6 months
  This outcome will be assessed by means of two specific questionaries
Denture quality (assessed by means of a clinical examination according to a specific form) | 3 months
  This outcome will be assessed by means of a clinical examination according to a specific form
Masticatory performance (assessed by means of a colorimetric method based on an artificial test food) | 6 months
  This outcome will be assessed by means of a colorimetric method based on an artificial test food

CONTACTS AND LOCATIONS:
Overall Officials: Romulo R Regis, DDS, PhD, Principal Investigator — romuloregis@hotmail.com
Locations (1):
- Dental School of Federal University of Ceara, Fortaleza, Ceará, Brazil

REFERENCES:
- [Background] Kawai Y, Murakami H, Shariati B, Klemetti E, Blomfield JV, Billette L, Lund JP, Feine JS. Do traditional techniques produce better conventional complete dentures than simplified techniques? J Dent. 2005 Sep;33(8):659-68. doi: 10.1016/j.jdent.2005.01.005. PMID 16139697
- [Background] Kawai Y, Murakami H, Takanashi Y, Lund JP, Feine JS. Efficient resource use in simplified complete denture fabrication. J Prosthodont. 2010 Oct;19(7):512-6. doi: 10.1111/j.1532-849X.2010.00628.x. Epub 2010 Aug 16. PMID 20723019
- [Background] Cunha TR, Della Vecchia MP, Regis RR, Ribeiro AB, Muglia VA, Mestriner W Jr, de Souza RF. A randomised trial on simplified and conventional methods for complete denture fabrication: masticatory performance and ability. J Dent. 2013 Feb;41(2):133-42. doi: 10.1016/j.jdent.2012.09.008. Epub 2012 Sep 19. PMID 23000525
- [Background] Regis RR, Cunha TR, Della Vecchia MP, Ribeiro AB, Silva-Lovato CH, de Souza RF. A randomised trial of a simplified method for complete denture fabrication: patient perception and quality. J Oral Rehabil. 2013 Jul;40(7):535-45. doi: 10.1111/joor.12063. Epub 2013 May 12. PMID 23663152
- [Background] Vecchia MP, Regis RR, Cunha TR, de Andrade IM, da Matta JC, de Souza RF. A randomized trial on simplified and conventional methods for complete denture fabrication: cost analysis. J Prosthodont. 2014 Apr;23(3):182-91. doi: 10.1111/jopr.12090. Epub 2013 Jul 26. PMID 23890072
- [Background] Omar R, Al-Tarakemah Y, Akbar J, Al-Awadhi S, Behbehani Y, Lamontagne P. Influence of procedural variations during the laboratory phase of complete denture fabrication on patient satisfaction and denture quality. J Dent. 2013 Oct;41(10):852-60. doi: 10.1016/j.jdent.2013.07.013. Epub 2013 Aug 1. PMID 23911602
- [Background] Nunez MC, Silva DC, Barcelos BA, Leles CR. Patient satisfaction and oral health-related quality of life after treatment with traditional and simplified protocols for complete denture construction. Gerodontology. 2015 Dec;32(4):247-53. doi: 10.1111/ger.12078. Epub 2013 Oct 21. PMID 24147575
- [Derived] Albuquerque IS, Freitas-Pontes KM, de Souza RF, Negreiros WA, Ramos MB, Peixoto RF, Regis RR. Is a two-step impression mandatory for complete denture fabrication on the severely resorbed mandible? A randomized trial on mastication, patient satisfaction and adjustments. J Dent. 2020 Aug;99:103357. doi: 10.1016/j.jdent.2020.103357. Epub 2020 May 8. PMID 32437857
- [Derived] Albuquerque IS, Regis RR, de Souza RF, Gurgel KF, Silva PG, Pinto-Fiamengui LMS, Freitas-Pontes KM. Is a two-step impression mandatory for complete denture fabrication on the severely resorbed mandible? A randomized trial on patient perception and denture quality. J Dent. 2020 Jul;98:103356. doi: 10.1016/j.jdent.2020.103356. Epub 2020 May 5. PMID 32380132